CLINICAL TRIAL: NCT04268485
Title: Longitudinal Changes in Serum KL-6 Levels in Idiopathic Pulmonary Fibrosis (LOCK-IPF)
Brief Title: Longitudinal Changes in Serum KL-6 in IPF
Acronym: LOCK-IPF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: ManchesterUNHS
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: KL-6; Krebs von den Lungen-6; Biomarker
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Medullary cystic kidney disease 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples taken on four separate visits over 12 months. Samples tested for KL-6 level onyl
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IPF patients: Patients with an MDT diagnosis of idiopathic pulmonary fibrosis. Patients will be observed over a 12 month period and have serial serum samples taken for KL-6 level.
  Interventions: Diagnostic Test: Serum KL-6 level

INTERVENTIONS:
Diagnostic Test: Serum KL-6 level — Serum blood biomarker which has been shown to be of interest in idiopathic pulmonary fibrosis

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a chronic lung disease with a poor prognosis. More accurate tests to predict disease progression and response to treatment are required.

Krebs von den Lungen-6 (KL-6) is a blood marker associated with IPF. Results from previous studies have shown that levels of KL-6 are higher in patients with IPF compared to people without the disease. In addition, it is not clear what impact treatment has on KL-6 levels, and whether this could help us to monitor how effective treatment for IPF is.

The investigators plan to perform a study in which KL-6 levels in the blood of patients with a new diagnosis of IPF are measured at baseline, 3, 6 and 12 months to look for and changes in the levels of KL-6 in the blood.

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis (IPF) is a chronic lung disease with a poor prognosis. Effective treatment which slows the progression of IPF has recently become available however, it is costly and at present is limited to patients who meet specific criteria based on their breathing tests. The breathing tests currently available to monitor progression of the disease are not always reliable and do not predict which patients will respond to treatment. More accurate tests to predict disease progression and response to treatment are required.

Krebs von den Lungen-6 (KL-6) is a blood marker associated with IPF. Results from previous studies have shown that levels of KL-6 are higher in patients with IPF compared to people without the disease. The majority of studies using KL-6 in IPF have taken place in Japan and there is limited evidence of how useful it is in a European population. In addition, it is not clear what impact treatment has on KL-6 levels, and whether this could help us to monitor how effective treatment for IPF is.

The investigators plan to perform a study in which KL-6 levels in the blood of patients with a new diagnosis of IPF are measured at baseline, 3, 6 and 12 months to look for and changes in the levels of KL-6 in the blood

The objective of this study is to assess changes in serum KL-6 levels in patients with IPF over a 12-month period and assess if this correlates with changes in lung function and if KL-6 levels change in response to treatment with antifibrotic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Multi-disciplinary team (MDT) diagnosis of idiopathic pulmonary fibrosis as per international consensus guidelines

Exclusion criteria

* Significant respiratory co-morbidity (i.e. where the major respiratory diagnosis is not IPF)
* FEV1/FVC ratio < 70% on full lung function testing
* Current smoker (within 4 week of enrollment)
* Received treatment for acute lower respiratory tract infection with last 4 weeks
* Use of long-term (greater than 4 weeks) oral corticosteroids or immunosuppression within 4 weeks of enrolment
* Current participation in a double-blind placebo-controlled pharmaceutical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an MDT diagnosis of idiopathic pulmonary fibrosis attending routine follow-up care
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Serum KL-6 level | 12 months
  Change in serum KL-6 level between baseline and 12 months

SECONDARY OUTCOMES:
Serum KL-6 level at 3, 6 months | 3 and 6 months
  Change in serum KL-6 at 3 and 6 months compared to baseline
KL-6 forced vital capacity (FVC) correlation | 3, 6 and12 months
  Correlation of KL-6 and FVC change at 3, 6 and 12 months
KL-6 diffusion capacity (DLCO) | 3, 6 and12 months
  Correlation of KL-6 and DLCO change at 3, 6 and 12 months
KL-6 symptoms | 3, 6 and12 months
  Correlation of KL-6 and symptom scores at 3, 6 and 12 months
KL-6 antifibrotics | 12 months
  Change in KL-6 levels in response to antifibrotic therapy
KL-6 Gender Age and Physiology (GAP) stage | At baseline
  Differences in KL-6 levels between Gender Age Physiology (GAP) stage at baseline
KL-6 CPI | At baseline
  Correlation between KL-6 levels and Composite Physiology Index (CPI)
KL-6 CT pattern | At baseline
  Difference in KL-6 levels between patients with indeterminate, probable and definite usual interstitial pneumonia pattern (UIP) on HRCT

CONTACTS AND LOCATIONS:
Overall Officials: Conal Hayton, Principal Investigator — Manchester University NHS Foundation Trust
Locations (1):
- Manchester University hospitals NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No